CLINICAL TRIAL: NCT01235455
Title: Portuguese BetaPlus Survey - Observational Study to Assess Drug Adherence in Patients With Multiple Sclerosis (MS) After Conversion to Betaferon by Using Elements of the BetaPlus Program
Brief Title: Portuguese Observational Survey to Assess Drug Adherence in Patients With Multiple Sclerosis After Conversion to Betaferon by Using Elements of the BetaPlus Program - Nurse Support, Auto-injectors
Acronym: POR-BetaPlus
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Portugal SA
Other Study IDs: 14235; BF0710PT (Other: Company internal)
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS); Secondary Progressive Multiple Sclerosis (SPMS)
Keywords: Multiple Sclerosis; Adherence; Interferon beta-1b; Coping styles
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — 250 µg, sub-cutaneously, on alternate days

SUMMARY:
This is an observational survey to assess the factors that influence adherence to Betaferon therapy in multiple sclerosis patients using elements of the BetaPlus support program, including the nurse support and auto-injectors. The patients were evaluated under normal clinical practice and were asked to fill out the quality of life FAMS questionnaire, Coping processes (WCQ) and depression questionnaire CES-D.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS (RRMS) or secondary-progressive MS (SPMS)
* Previous treatment with disease modifying drugs
* Adjustment of disease modifying treatment necessary at the discretion of the investigator
* Switch to Betaferon at least 1 month but not longer than 3 months prior to inclusion

Exclusion Criteria:

* Patients not fulfilling the indications in the local prescribing information
* Refusal to sign inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RRMS or SPMS attending an hospital outpatient MS clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-08; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Identification of reasons why patients are switched from other disease modifying drugs to Betaferon due to perceived lack of efficacy, adverse events, poor compliance, and others. | After 2 years
Assessment of factors predictive of non-adherence to disease modifying drugs such as demographic data, course of disease, drug history, patients characteristics, history of poor compliance to prior therapy or others. | After 2 years

SECONDARY OUTCOMES:
Assessment of impact of supportive elements of the BetaPlus Program like nurse support, auto-injector, website, etc on treatment adherence. | After 2 years
Evaluation of impact of Betaferon treatment on health related quality of life using the Functional Assessment of Multiple Sclerosis Questionnaire - FAMS. | After 2 years
Assessment of coping processes by applying the Ways of Coping Questionnaire. | After 2 years
Measurement of safety of Betaferon by assessing the number of participants with adverse events and severe adverse events. Classification by MedDRA category. | After 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Portugal